CLINICAL TRIAL: NCT02072876
Title: Asymptomatic Intracranial Atherosclerotic Disease: Prevalence, Clinical and Lifestyle Determinants in Urban Pakistan
Brief Title: Asymptomatic Intracranial Atherosclerotic Disease in Pakistanis
Acronym: AICAD
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Ayeesha Kamran Kamal, Associate Professor Neurology,Director Stroke Fellowship Program, Aga Khan University
Other Study IDs: 5D43TW008660-03 (NIH)
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Intracranial Atherosclerosis
Keywords: Stroke; Asymptomatic Intracranial Atherosclerotic Disease; Lifestyle and socio-economic risk factors; Clinical predictors
MeSH Terms: conditions — Intracranial Arteriosclerosis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Asymptomatic ICAD on MRI Absent: Those who test negative on QVSFS, Questionnaire to Verify Stroke Free Status, and do not have ICAD on MRI. They are clinically and biologically free of disease.
- Asymptomatic ICAD Present on MRI: Those who are negative for Stroke Symptoms on QVSFS, Questionnaire to Verify Stroke Free Status, yet have evidence of ICAD on MRI

SUMMARY:
The incidence of stroke has increased by 100% in the last four decades in developing countries like Pakistan. Intracranial atherosclerotic disease (ICAD) is the most frequent causative subtype of ischemic stroke in the world including Pakistan. ICAD is progressive narrowing of the arteries at the base of the brain due to atherosclerosis. After a stroke from ICAD, recurrence rate is highest in any sub-type of stroke, up to 28% with limited therapeutic options. Therefore, it is imperative to delineate the determinants of asymptomatic ICAD prior to stroke. Investigators hypothesized that there is at least a 20% difference in the proportion of clinical, life-style (dietary, physical activity, obesity, smoking and stress/depression), and socio-economic predictors of asymptomatic ICAD than those with no ICAD.

DETAILED DESCRIPTION:
Stroke is a major emerging cause of adult disability and the 3rd leading non-communicable cause of mortality in the world . With half of the world's population living in Asia, stroke epidemiology and its risk factor determination is important globally. The changes in population demographics and continuing industrialization in Asia have also led to a change in the epidemiology of stroke sub-types . Among the ischemic stroke sub-types, Intracranial Atherosclerotic disease is now emerging as the most prevalent vascular cause of stroke with high prevalence in Asian, African and Hispanic individuals .

Patients with ICAD are at a significant risk for recurrent stroke, with a risk as high as 25% in the first two years . Rate of recurrent stroke also varies by the location of the affected artery. Risk factor management is extremely important for the primary and secondary prevention of stroke in Asia as it is in Western countries. With the changing demographics and relatively fewer cost effective treatment modalities available, particularly for resource poor countries like Pakistan, it is imperative to delineate the clinical as well as lifestyle risk factors at an earlier asymptomatic stage to prevent future life-threatening consequences.

Therefore the primary objective of this study is to determine the clinical, lifestyle, dietary and psycho-social determinants of asymptomatic Intracranial Atherosclerotic disease (ICAD) and its other associated Brain MRI findings namely brain volume reduction, silent brain infarcts, and peri-ventricular hyper intensities in clinically normal adults with ICAD on MRI Brain.

ELIGIBILITY:
Inclusion Criteria:

* Adult Pakistani men and women ≥ 18years getting MRI brain for any indication other than stroke.
* Permanent residents of Pakistan for at least 1 year.
* No prior history of stroke which was confirmed by screening with Questionnaire for verifying stroke free status (QVSFS).
* Able to give written informed consent.

Exclusion Criteria:

* QVSFS +ve.
* Severe disability, life expectancy less than 6 months at enrollment.
* Patients in whom MRI prolongation for 5 minutes can be harmful for the patient (Anesthesia, claustrophobia, sedation etc.).
* Any clear contraindications to MRI, like pacemakers, metallic valves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study recruited all adult Pakistani patients ≥ 18 yrs., with no previous clinical history of stroke, (negative on QVSFS; Questionnaire to Verify Stroke Free Status), presenting to the two tertiary care centers for MRI Brain for indications other than stroke.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Distribution and Degree of Asymptomatic Intracranial Stenosis | MRA , Once , Over One Year
  This was defined as any artery (Internal Carotid Artery ICA, Middle Cerebral Artery MCA,Anterior Cerebral Artery ACA,Posterior Cerebral Artery PCA, Basilar Artery BA, and Vertebral Artery VA) having >25% stenosis on MRA. An internationally standardized ( WASID) equation was used to calculate the degree of stenosis.
  Percent stenosis= [1- (Dstenosis/D normal)*100], where D Stenosis is the diameter of the artery at the site of the most severe stenosis, and D normal= diameter of the proximal normal artery.

SECONDARY OUTCOMES:
Associated Brain MRI Findings with Intracranial Stenosis | MRA Once , Over One Year
  Brain volume reduction, Central and Peripheral Atrophy Periventricular Lucencies Silent Brain Infarcts

CONTACTS AND LOCATIONS:
Overall Officials: Ayeesha K Kamal, MBBS, Principal Investigator — Aga Khan University
Locations (2):
- Pakistan (2):
  - Aga Khan University, Karachi, Sindh
  - Akuh,Duhs, Karachi, Sindh

REFERENCES:
- [Derived] Kamal AK, Majeed F, Pasha O, Islam M, Azam I, Ilyas MS, Hussain M, Masood K, Ahmed B, Nazir S, Sajjad Z, Kasner SE. Study protocol: asymptomatic intracranial atherosclerotic disease in pakistanis. J Vasc Interv Neurol. 2015 Feb;8(1):27-35. PMID 25825629
- [Derived] Kamal AK, Majeed F, Pasha O, Rehman H, Islam M, Azam I, Ilyas MS, Hussain M, Masood K, Ahmed B, Nazir S, Sajjad Z, Kasner SE. Clinical, lifestyle, socioeconomic determinants and rate of asymptomatic intracranial atherosclerosis in stroke free Pakistanis. BMC Neurol. 2014 Aug 15;14:155. doi: 10.1186/s12883-014-0155-6. PMID 25124284